CLINICAL TRIAL: NCT00236639
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter, Parallel Group, Dose-Response Study to Assess the Efficacy and Safety of Topiramate in the Treatment of Patients With Obesity
Brief Title: A Study on Efficacy and Safety of Topiramate in the Treatment of Patients With Obesity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR003721
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2010-04-28 (Estimated); Status verified 2010-04

CONDITIONS: Obesity
Keywords: Obesity; Hypertension; Hyperlipidemia; Type 2 Diabetes Mellitus; Body Mass Index
MeSH Terms: conditions — Obesity; Hypertension; Hyperlipidemias; Diabetes Mellitus, Type 2 | interventions — Topiramate

INTERVENTIONS:
Drug: topiramate

SUMMARY:
The purpose of this study is to compare the efficacy and safety of topiramate (96, 192, and 256mg daily) with placebo in long-term treatment of obesity.

DETAILED DESCRIPTION:
Topiramate is not approved for the treatment of obesity. This double-blind, placebo-controlled study assesses long-term effectiveness and safety of topiramate in patients with obesity. After completing 6 weeks of run-in phase (a single-blind placebo-treatment phase during which patients begin non-pharmacological therapy), patients will be randomized to receive either topiramate or placebo. Topiramate group will receive 16mg of topiramate and the dose will be titrated over 8 weeks. Patients will then receive two years of treatment. Effectiveness will be evaluated by body weight, Body Mass Index (BMI), anthropometric measurements (waist circumference, hip circumference, waist/hip ratio), fasting lipid profile, fasting plasma glucose, HbA1c, fasting uric acid, fasting insulin, blood pressures, body fat compositions, mass of left ventricle of the heart (as measured by echocardiography), and Health Related Quality of Life scores. Safety evaluation (incidence of adverse events, laboratory tests, electrocardiogram, vital signs) will be performed throughout the study. The study hypothesis is that topiramate will be effective in achieving and maintaining weight reduction in obese patients. During the initial 8 weeks, the doses of topiramate or placebo will be gradually increased to the target dose (either 96mg, 192mg, or 256mg daily by mouth) and the doses will be maintained for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) >= 30 and < 50
* BMI >= 27 and < 50 if patient has controlled hypertension or abnormal blood lipids
* Stable weight
* Female patients must be postmenopausal for at least 1 year, surgically incapable of childbearing, practicing abstinence, or practicing an acceptable method of contraception (requires negative pregnancy test)

Exclusion Criteria:

* Known contraindication, or hypersensitivity to topiramate
* A diagnosis of diabetes (except those diagnosed during the enrollment if no medications are needed)
* History or evidence of clinically significant liver, disease, cardiovascular disease, uncontrolled hypertension or high thyroid levels
* History of obesity with known cause
* History of weight loss surgery or liposuction
* History of malignancy within last 5 years

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1293 (Actual)
Dates: Start 2000-07; Study Completion 2002-06 (Actual)

PRIMARY OUTCOMES:
The percent change in body weight from the baseline (randomization) to Week 60 (after one year of maintenance therapy).

SECONDARY OUTCOMES:
Changes from either baseline to Week 60 and/or Week 112, or enrollment to Week 60 and/or Week 112 in absolute body weight, Body Mass Index (BMI), body measurements, fasting lipid profile.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Wilding J, Van Gaal L, Rissanen A, Vercruysse F, Fitchet M; OBES-002 Study Group. A randomized double-blind placebo-controlled study of the long-term efficacy and safety of topiramate in the treatment of obese subjects. Int J Obes Relat Metab Disord. 2004 Nov;28(11):1399-410. doi: 10.1038/sj.ijo.0802783. PMID 15486569